CLINICAL TRIAL: NCT06058689
Title: A Pilot, Open-label, Randomized, Two-Way Crossover, Single-Dose Bioequivalence Study of Pomalidomide Under Fasting Condition in Indian Healthy Volunteers
Brief Title: A Pilot Bioequivalence Study of Pomalidomide
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Megalabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Pomalidomide
Record Dates: First submitted 2023-09-15; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Bioequivalence Study
MeSH Terms: interventions — pomalidomide

STUDY DESIGN:
Intervention Model Description: An open label, balanced, randomized, two treatments, two sequences, two periods, single dose, crossover, bioequivalence study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pomalidomide Test (Experimental): Pomalidomide 4 MG Oral Capsule per os,1 capsule per period
  Interventions: Drug: Pomalidomide 4 MG Oral Capsule
- Pomalidomide Reference (Experimental): Pomalidomide 4 MG Oral Capsule (Pomalyst) per os,1 capsule per period
  Interventions: Drug: Pomalidomide 4 MG Oral Capsule

INTERVENTIONS:
Drug: Pomalidomide 4 MG Oral Capsule — A single dose of 4 mg Pomalidomide per os, capsule, 4 mg, per period
  Other Names: Pomalyst, Pomalidomide Megalabs

SUMMARY:
Pilot bioequivalence trial of two pomalidomide formulations consisting in 4 mg oral capsules.

DETAILED DESCRIPTION:
An open label, balanced, randomized, two treatments, two sequences, two periods, single dose, crossover assignment, bioequivalence study of Pomalidomide 4 mg Capsules of Mega Labs S.A and Pomalyst® (Pomalidomide) 4 mg capsules of Celgene International SARL, Boudry, Switzerland in healthy, adult, human male subjects under fasting condition.

ELIGIBILITY:
Inclusion Criteria:

Healthy male literate volunteers of 18 to 45 years with BMI of 18.50 - 29.99 Kg/m2 and weight > 50 Kg.

Healthy volunteers as evaluated by medical history, vitals and general clinical examination.

Normal or clinically insignificant biochemical, hematological, urine and serology parameters.

Normal or clinically insignificant ECG. Negative urine test for drugs of abuse, alcohol breath analysis. Volunteers who are willing to use acceptable methods of contraception. Volunteers who can give written informed consent and communicate effectively.

Exclusion Criteria:

History of any major surgical procedure in the past 03 months. History of any clinically significant cardiac, gastrointestinal, respiratory, hepatic, renal, endocrine, neurological, metabolic, psychiatric and hematological disorders.

History of chronic alcoholism/ chronic smoking/ drug of abuse. Volunteers with known hypersensitivity to Pomalidomide or any of the excipients.

History of consumption of tobacco containing products within 48 hours prior to proposed time of dosing Volunteer who are positive for hepatitis B surface antigen, anti-hepatitis C antibody, treponemal antibodies and human immunodeficiency virus (HIV 1&2) antibodies.

Present or past history of intake of drugs or any prescription drug or over the counter (OTC) drugs within 14 days which potentially modify kinetics / dynamics of Pomalidomide or any other medication judged to be clinically significant by the investigator.

History of consumption of grapefruit and/or its products within 10 days prior to the start of study.

Volunteer who had participated in any other clinical study or who had bled during the last 03 months before check-in.

History of consumption of one or more of the below, 48 hours prior to dosing: Xanthine containing food or drinks such as cola, chocolate, coffee or tea, citrus fruits or items (lime, lemon and orange), alcohol and any other food/beverage known to have interactions as deemed by the investigator Volunteers who are dysphagic

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2024-11-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Cmax | Day 1, Day 2, Day 3 of cycle 1, Day 8, Day 9, Day 10 of cycle 2.
  Peak Plasma Concentration (Cmax). T/R of Cmax R within 80-125% for IC 90% vs the Comparator; also to generate pharmacokinetic data that can be used to design a pivotal bioequivalence study.
AUC0-t | Day 1, Day 2, Day 3 of cycle 1, Day 8, Day 9, Day 10 of cycle 2. 90% CI of T/R within 80-125%
  Area under the plasma concentration versus time curve from 0 to the last measurable concentration (AUC0-t). T/R of AUC 0-t within 80-125% for 90% CI vs the Comparator.
AUC0-inf | Day 1, Day 2, Day 3 of cycle 1, Day 8, Day 9, Day 10 of cycle 2. 90% CI of T/R within 80-125%
  Area under the plasma concentration versus time curve from 0 to the last measurable concentration (AUC0-t). T/R of AUC 0-t within 80-125% for 90% CI vs the Comparator.

CONTACTS AND LOCATIONS:
Overall Officials: M. Gowtham, MD, Principal Investigator — Azidus Laboratories
Locations (1):
- Azidus Laboratories, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No